CLINICAL TRIAL: NCT04609020
Title: Prospective, Multi-site Study to Evaluate Subject Satisfaction With Facial Appearance Overall and the Aesthetic and Psychosocial Impact of Combined Facial Treatment
Brief Title: Study to Evaluate Subject Satisfaction With Facial Appearance and Impact of Combined Facial Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-FAS-0580
Record Dates: First submitted 2020-10-06; First posted 2020-10-30 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Facial Rhytides; Skin Folds; Loss of Volume and Skin Quality
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HArmonyCA, Juvederm, BOTOX (Experimental): All treatments will be administered according to the respective label and according to an agreed upon treatment plan between the subject and Health Care Provider. If required: HarmonyCA Lidocaine will be administered at Visit 1, Juvéderm filler injections (JUVÉDERM VOLBELLA with Lidocaine, and/or JUVÉDERM VOLIFT with Lidocaine, and/or JUVÉDERM VOLUMA with Lidocaine, and/or JUVÉDERM VOLITE with Lidocaine and/or JUVÉDERM VOLUX with Lidocaine) will be administered at Visit 3, BOTOX will be administered at Visit 5. Touch-ups may be performed as required by subject's treatment plan after each study visit.
  Interventions: Device: JUVÉDERM; Drug: BOTOX; Device: HArmonyCA Lidocaine

INTERVENTIONS:
Device: JUVÉDERM — JUVÉDERM VOLBELLA with Lidocaine Treatment of any fine lines and medium-sized skin depressions. Can also be used for enhancement and pouting of the lips to correct structural defects such as asymmetry, contour deformities, volume loss. JUVÉDERM VOLIFT with Lidocaine Intended for the treatment of any deep skin depressions due to conditions such as premature aging. Can also be used for face contouring and volume restoration to correct facial structural defects such as asymmetry, contour deformities, volume loss in the lips, cheeks, chin, lower face. JUVÉDERM VOLUMA with Lidocaine Intended to restore volume of the face JUVÉDERM VOLITE with Lidocaine Intended for treatment, by filling, of superficial cutaneous depressions such as fine lines and for additional improvement of skin quality attributes such as hydration and elasticity. JUVÉDERM VOLUX with Lidocaine Intended to restore and generate facial volume in chin and mandible areas
Drug: BOTOX — Indicated for the treatment of hyperkinetic facial lines.
Device: HArmonyCA Lidocaine — HArmonyCa Lidocaine injectable gel is a dermal filler intended for facial soft tissue augmentation.

SUMMARY:
The primary objective of this study is to quantify the psychological, social, and emotional impact of comprehensive aesthetic treatment with a portfolio of the Sponsor's products by measuring the change in subject's satisfaction with facial appearance from baseline (before any treatment) to the final study visit

ELIGIBILITY:
Inclusion Criteria:

* Accept the obligation not to receive any other facial procedures or treatments at any time during the study that are not related to the study
* Women of childbearing potential must have a negative urine pregnancy test before each injectable treatment and practice a reliable method of contraception throughout the study
* Willing to avoid direct and prolonged sun exposure to the facial skin, which includes tanning beds, for the duration of the study
* Must qualify to receive BOTOX treatments, in at least one area, as per the approved Product Monograph including treatment of hyperkinetic lines for the glabellar, crow's feet, and forehead lines:

  * Glabellar injection: glabellar rhytides characterized as moderate or severe during maximum muscle contraction on the evaluation of the facial wrinkle scale (FWS)
  * CFLs characterized as 2 (moderate) or 3 (severe) during maximum smile on the evaluation of the FWS
  * Forehead lines (FHLs) of moderate to 3 severe rating at maximum eyebrow elevation as assessed using the FWS

Exclusion Criteria:

* Body mass index (BMI) > 30 kg/m2
* Known allergy or sensitivity to the study products or their components
* Pregnant, lactating, or planning to become pregnant at any time during the study
* Received BOTOX or treatment with any other botulinum toxin product for any condition within 6 months before enrollment
* Received (or is planning to receive) anti-coagulation, antiplatelet or thrombolytic medications (e.g., warfarin) or other substances known to increase coagulation time from 10 days prior to injection and up to 3 days post-injection
* Undergone plastic surgery of the face and/or neck, tissue grafting, or tissue augmentation with silicone, fat, or other permanent dermal fillers, or be planning to undergo any of these procedures at any time during the study
* Has undergone temporary or semi-permanent facial or neck dermal filler treatment (e.g., hyaluronic acid, calcium hydroxylapatite, poly-L-lactic acid) within 12 months before enrollment
* Received mesotherapy, skin resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or non-ablative procedures) in the face or neck within 6 months prior to study enrollment
* Marked facial asymmetry, brow or eyelid ptosis, excessive dermatochalasis, deep dermal scarring, thick sebaceous skin, or an inability to substantially lessen the resting GLs and CFLs/facial rhytides by physically spreading them apart
* Lip tattoos, facial hair or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
* At any proposed injection site, presence of inflammation, infection at any injection site or systemic infection (study entry may be postponed until one week following recovery), noticeable acne scarring, cancerous or pre-cancerous lesion, or unhealed wound or have undergone radiation treatment in the area to be treated
* Received any investigational product within 60 days prior to study enrollment or planning to participate in another investigation during the course of this study
* Current use of oral corticosteroids
* Current use of nonsteroidal anti-inflammatory drugs (NSAIDs) (e.g., aspirin, ibuprofen), from 10 days prior to injection up to 3 days post-injection
* Prescription topical retinoid therapy and/or topical hormone cream applied to the face, for potential subjects who have not been on a consistent dose regimen for at least 6 months prior to enrollment and who are unable to maintain regimen for the study
* Systemic retinoid therapy within one year prior to study enrollment
* History or current symptoms of dysphagia
* Medical condition that may increase the risk of exposure to botulinum toxin including diagnosed myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function
* Profound atrophy/excessive weakness of muscles in target areas of injection
* History of facial nerve palsy
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study treatment)
* Very thin skin in the mid-facial region
* Tendency to accumulate fluid in the lower eyelids, or large infraorbital fat pads, i.e., significant convexity or projection from the infraorbital fat pads
* Mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or human immunodeficiency virus-related disease
* Undergone oral surgery or other dental procedures (e.g., tooth extraction, orthodontia, or implantation) within 30 days prior to enrollment or be planning to undergo any of these procedures during the study
* Subjects with neuromuscular disorders including generalized muscle weakness, diplopia, ptosis, dysphonia, dysarthria, severe dysphagia, and respiratory compromise
* Subjects with a history of allergies

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (6):
- Brazil (6):
  - Hospital Regional da Asa Norte - Brasilia /ID# 239161, Brasília, Federal District
  - Hospital do Servidor Publico Municipal - Sao Paulo /ID# 239165, Niterói, Rio de Janeiro
  - Universidade de Sao Paulo - Sao Paulo /ID# 239163, Rio de Janeiro
  - Dermick Clinica de Dermatologia - Niteroi/Rio de Janeiro /ID# 239166, São Paulo
  - BRAVOMED Dermatology - Rio de Janeiro /ID# 239160, São Paulo
  - Universidade Federal de Sao Paulo - Sao Paulo /ID# 239156, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Groups:
- HArmonyCA: All treatments will be administered according to the respective label and according to an agreed upon treatment plan between the subject and Health Care Provider. If required: HarmonyCA Lidocaine will be administered at Visit 1, Juvéderm filler injections (JUVÉDERM VOLBELLA with Lidocaine, and/or JUVÉDERM VOLIFT with Lidocaine, and/or JUVÉDERM VOLUMA with Lidocaine, and/or JUVÉDERM VOLITE with Lidocaine and/or JUVÉDERM VOLUX with Lidocaine) will be administered at Visit 3, BOTOX will be administered at Visit 5. Touch-ups may be performed as required by subject's treatment plan after each study visit.
  Device: HArmonyCa Lidocaine injectable gel is a dermal filler intended for facial soft tissue augmentation.
Period: Overall Study
Arm/Group | HArmonyCA
Started (A total of 65 subjects were screened and 64 subjects were enrolled in the study. There was 1 screen failure due to "other: pause in study recruitment".) | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HArmonyCA
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Rasch-transformed Score of the FACE-Q Satisfaction With Facial Appearance Scale.
Description: The FACE-Q questionnaire focuses on patient's satisfaction with facial appearance at the final study visit compared to before starting study treatment and is a 10- item questionnaire. Overall scores range from 0 to 100 with higher scores representing higher satisfaction.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
units on a scale | 46.6 (23.61)
Statistical Analysis 1: Comparison: HArmonyCA; Test type: Superiority; p < 0.0001, t-test, 1 sided — P-value is calculated based on 1-sided t-test or Wilcoxon signed-rank test (if the normality assumption is not met) at 0.025 significance level; Mean Difference (Final Values) = 46.6, 97.5% CI 1-sided [lower limit 40.58], Standard Deviation 23.61

2. Secondary Outcome: Change From Baseline in the FACE-Q Aging Appraisal
Description: The FACE-Q questionnaire is a 7-item questionnaire with overall scores that range from 0 to 100 and higher scores reflecting a better outcome.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
units on a scale | 35.3 (22.36)
Statistical Analysis 1: Comparison: HArmonyCA; Test type: Superiority; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 35.3, 97.5% CI 1-sided [lower limit 29.61], Standard Deviation 22.36

3. Secondary Outcome: Change From Baseline in the Rasch-transformed Score of the FACE-Q Psychological Function Scale
Description: The FACE-Q questionnaire is a 10-item questionnaire with overall scores that range from 0 to 100 and higher scores reflecting a better outcome.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
units on a scale | 27.6 (23.23)
Statistical Analysis 1: Comparison: HArmonyCA; Test type: Superiority; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 27.6, 97.5% CI 1-sided [lower limit 21.50], Standard Deviation 23.23

4. Secondary Outcome: Change From Baseline in the Rasch-transformed Score of the FACE-Q Social Function Scale
Description: The FACE-Q questionnaire is a 8-item questionnaire with overall scores that range from 0 to 100 and higher scores reflecting a better outcome.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
units on a scale | 22.9 (20.56)
Statistical Analysis 1: Comparison: HArmonyCA; Test type: Superiority; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 22.9, 97.5% CI 1-sided [lower limit 17.65], Standard Deviation 20.56

5. Secondary Outcome: Change From Baseline in the Rasch-transformed Score of the FACE-Q Satisfaction With Skin
Description: The FACE-Q questionnaire is a 12- item questionnaire. Overall scores range from 0 to 100 with higher scores representing higher satisfaction.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
units on a scale | 43.1 (22.25)
Statistical Analysis 1: Comparison: HArmonyCA; Test type: Superiority; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 43.1, 97.5% CI 1-sided [lower limit 37.48], Standard Deviation 22.25

6. Secondary Outcome: Change From Baseline Self-Perception of Age
Description: Subject's assessment of self-perception of age as measured by SPA. Subject's selected one of 3 options based on how they felt their facial appearance looked compared to their age on the day they completed the assessment, writing in the number of years when appropriate.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable Population
Measure: Median (Full Range); unit: years
Arm/Group | HArmonyCA
Number analyzed (Participants) | 15
years
  I look ___ years younger | 3.0 [0 to 13]
  I look ___ years older | 0 [0 to 0]

7. Secondary Outcome: Investigator's Assessment Using Global Aesthetic Improvement Scale (GAIS)
Description: Five point ordinal scale measuring the change in facial aesthetic improvement from -2 (Much Worse) to 2 (Much Improved) assessed by the Investigator.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
Participants
  Much Improved | 47
  Improved | 15
  No Change | 0
  Worse | 0
  Much Worse | 0

8. Secondary Outcome: Subject's Assessment Using Global Aesthetic Improvement Scale (GAIS)
Description: Five point ordinal scale measuring the change in facial aesthetic improvement from -2 (Much Worse) to 2 (Much Improved) assessed by the subject.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
Participants
  Much Improved | 51
  Improved | 11
  No Change | 0
  Worse | 0
  Much Worse | 0

9. Secondary Outcome: Change From Baseline to End of Study of Periorbital Aesthetic Appearance Questionnaire (PAAQ)
Description: Questionnaire evaluating the subject's overall eye appearance from 0 (Never) to 4 (All of the Time) for each of the 9 items. All items were transformed to a scale from 0 (no negative impact) to 100 (high negative impact).
  Total transformed score is based on 9 individual items each item has a range of 0 to 4, the transformed score ranges from 0 to 100.
  Psychological domain is based on the average of the sum of transformed scores of individual items 2, 4, 6, 7, and 8. Score will also range from 0 to 100 with same interpretation as the total transformed score.
  Appearance domain is based on the average of the sum of transformed scores of individual items 1, 3, and 5. Score will also range from 0 to 100 with same interpretation as the total transformed score.
  Coping domain is the transformed score of item 9. Score will also range from 0 to 100 with same interpretation as the total transformed score.
Time Frame: Visit 0 (Day 1) to Visit 7 (Up to approximately 5 months)
Population: Evaluable population
Measure: Median (Full Range); unit: units on a scale
Arm/Group | HArmonyCA
Number analyzed (Participants) | 62
units on a scale
  Change from Baseline Transformed Total Score | -40.3 [-86 to 39]
  Change from Baseline Psychological Domain | -40.0 [-90 to 45]
  Change from Baseline Appearance Domain | -45.8 [-100 to 42]
  Change from Baseline Coping Domain | -50.0 [-100 to 25]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 147 days for HArmonyCA.
Arm/Group | HArmonyCA
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 2/64
Other Adverse Events (participants affected / at risk) | 8/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HArmonyCA (N=64)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HArmonyCA (N=64)
PERIORBITAL OEDEMA (Eye disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
LIP OEDEMA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
INJECTION SITE BRUISING (General disorders) | 1 (1)
INJECTION SITE INDURATION (General disorders) | 1 (1)
INJECTION SITE NODULE (General disorders) | 1 (1)
INJECTION SITE OEDEMA (General disorders) | 2 (3)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
DENGUE FEVER (Infections and infestations) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT04609020/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT04609020/SAP_001.pdf